CLINICAL TRIAL: NCT05427045
Title: A Pilot Project for Multifidus Muscle Evaluation in Patients With Multiple Sclerosis and Back Pain
Brief Title: A Pilot Project for Multifidus Muscle Evaluation in Patients With Multiple Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Incomplete follow up, low enrollment
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 263068
Record Dates: First submitted 2022-05-23; First posted 2022-06-22 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis; Back Pain
MeSH Terms: conditions — Multiple Sclerosis; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Adult patients < 50 years old who have multiple sclerosis and back pain who are undergoing home exercise
  Interventions: Other: home - exercise program

INTERVENTIONS:
Other: home - exercise program — Home exercise program

SUMMARY:
This research study plans to evaluate if multifidus muscle dysfunction is associated with back pain in patients with Multiple Sclerosis (MS).

DETAILED DESCRIPTION:
Since the multifidus muscle helps to stabilize the lumbar spine, the investigators hope to learn if there is dysfunction and/or atrophy of this muscle in MS patients who also have back pain. The main objective is to study if it is possible to do a home-exercise program in patients with MS younger then 50 years old and who do not need any assistance to walk. Another objective is to further characterize the multifidus function in those patients. This will be by by measuring the size of muscle at the beginning and end of the study, and also by physical exam. As an exploratory aim, the investigators would like to evaluate the relation between compliance with the home-exercise program and the change in the size of the multifidus muscle and the change in pain.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis by an UAMS neuro-immunologist of relapsing-remitting MS or primary progressive MS or secondary progressive MS
* Age between 18 years old and 50 years old on consent
* Complain of low back pain or severe axial back pain
* English-speaking

Exclusion Criteria:

* Patients that also have the diagnosis of thoracic or lumbar radiculopathy or history of prior thoracic or lumbar spinal surgery.

Patients that are currently pregnant EDSS over 5.5 or less than 1.0 Patient younger than 18 years old or older than 50 years old Knee total extension of less than 100 degrees

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erika Santos Horta, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group
Started | 7
Completed | 1
Not Completed | 6

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Other: home - exercise program Home exercise program
Arm/Group | Intervention Group
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Study the Compliance of a Home-exercise Program in Patients With MS
Description: we will evaluate how many exercise sessions patients do at home versus what was purposed to the patient.
Time Frame: 6 months
Population: Patient never returned to Physical Therapy - no data was collected
Arm/Group | Intervention Group
Number analyzed (Participants) | 0

2. Secondary Outcome: Qualify the Multifidus Dysfunction in Patients With MS - Ultrasound
Description: evaluation of the change from baseline of a cross-section area of the multifidus muscle measured by ultrasound
Time Frame: 6 months
Population: No subject completed study- No data was collected as subject did not return for visit
Units Other Than Participants: Change on Cross section
Arm/Group | Intervention Group
Number analyzed (Participants) | 0
Number analyzed (Change on Cross section) | 0

3. Secondary Outcome: Qualify the Multifidus Dysfunction in Patients With MS - Physical Exam
Description: evaluation of the change from baseline of a cross-section area of the multifidus muscle measured by physical exam maneuvers
Time Frame: 6 months
Population: Subject never returned for PT- no data was collected
Arm/Group | Intervention Group
Number analyzed (Participants) | 0

4. Secondary Outcome: Correlation Between Compliance and Plain and Size of Muscle
Description: statistical analysis will be done to verify the relation between compliance with the home-exercise program and the change in the cross-section area of the multifidus muscle and the change in pain score using PROMIS scale
Time Frame: 6 months
Population: Subject never returned to clinic to complete pain score- No data was collected
Arm/Group | Intervention Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year from the time a subject was enrolled
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT05427045/Prot_SAP_000.pdf